CLINICAL TRIAL: NCT04431336
Title: Clinical Characters, Treatment and Prognosis of the Young Patient With Aortic Dissection or Aneurysm: A Prospective Observational Cohort Study
Brief Title: Young Patient With Aortic Dissection or Aneurysm: A Prospective Observational Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chinese Medical Association (Network)
Collaborators: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zaiping Jing, Professor, Chinese Medical Association
Other Study IDs: https://orcid.org/0000-0002-04
Record Dates: First submitted 2020-06-08; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Aortic Aneurysm and Dissection
MeSH Terms: conditions — Aortic Dissection | interventions — Movement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — To explore pathogenic genes 5m peripheral blood was extracted for whole genome sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- younger aortic dissection or aneurysm patients: this is an observation cohort study about younger aortic dissection or aneurysm patients without intervention.
  Interventions: Behavioral: movement

INTERVENTIONS:
Behavioral: movement — movement

SUMMARY:
Aortic dissection or aneurysm is unusual in young patients, and frequently associated with unusual presentations. However studies about this area is scarce. Besides, the treatment option is not clare. The prognosis of this cohort is also unclear.

The goal of this study was to better understand the characters, treatment option and prognosis of young patient with aortic dissection or aneurysm.

DETAILED DESCRIPTION:
To understand the clinical characteristics, treatment options and prognosis of aortic dissection or aneurysm in young people，the study plan will include young people younger (≤50 years) with aortic dissection or aneurysm from 2020.6. Then collect their clinical data and conduct follow-up studies, in order to understand younger aortic dissection or aneurysm patients.

ELIGIBILITY:
Inclusion Criteria:

* young patients with aortic dissection or aneurysm

Exclusion Criteria:

* Aortic dissection or aneurysm due to traumatic

Ages: 1 Year to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: young patients aged less than 50 years old and had aortic dissection or aneurysm
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-05 (Estimated); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical features of young aortic dissection and aneurysm patients | before December 2021
  Collecting clinical data, such as basic information, blood biochemical information and imaging informatio to describe the characteristics of young people.

CONTACTS AND LOCATIONS:
Overall Officials: Zaiping MD Jing, Professor, Principal Investigator — Vascular surgery, Changhai Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Januzzi JL, Isselbacher EM, Fattori R, Cooper JV, Smith DE, Fang J, Eagle KA, Mehta RH, Nienaber CA, Pape LA; International Registry of Aortic Dissection (IRAD). Characterizing the young patient with aortic dissection: results from the International Registry of Aortic Dissection (IRAD). J Am Coll Cardiol. 2004 Feb 18;43(4):665-9. doi: 10.1016/j.jacc.2003.08.054. PMID 14975480
- See also: Characterizing the young patient with aortic dissection: results from the International Registry of Aortic Dissection (IRAD). — https://pubmed.ncbi.nlm.nih.gov/14975480/?from_single_result=Characterizing+the+Young+Patient+With+Aortic+Dissection%3A+Results+From+the+International+Registry+of+Aortic+Dissection+%28IRAD%29&solr_messages=%7B%22messages%22%3A+%5B%22Custom+filter+IF%3A5-10+is+ignored+because+its+expression+exceeds+4000+characters.%22%2C+%22Custom+filter+IF%3A3-5+is+ignored+because+its+expression+exceeds+4000+characters.%22%2C+%22Custom+filter+IF%3A%3E10+is+ignored+because+its+expression+exceeds+4000+characters.%22%2C+%22Custom+filter+IF%3A2-3+is+ignored+because+its+expression+exceeds+4000+characters.%22%5D%7D